CLINICAL TRIAL: NCT02513615
Title: Epigenetic Determinants of Peritoneal Fibrosis
Status: Completed | Type: Observational
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Peter Margetts, Principle investigator, McMaster University
Other Study IDs: 14CECPDNA1006
Record Dates: First submitted 2015-07-30; First posted 2015-07-31 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Peritoneal Fibrosis
Keywords: Fibrosis; Peritoneal Dialysis; Epigenetics; Peritoneal membrane injury; Glucose exposure
MeSH Terms: conditions — Peritoneal Fibrosis; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A 15ml sample of PD fluid
Oversight: Data Monitoring Committee: No

SUMMARY:
Peritoneal dialysis (PD) is a type of kidney replacement therapy for patients with chronic kidney disease where the peritoneal membrane is used to filter the blood. Exposure to PD fluid results in scarring of the peritoneal membrane and increased blood vessel growth. This condition can progress even when peritoneal dialysis is stopped. Therefore, the investigators hypothesize glucose in the dialysis fluid may result in DNA modifications called epigenetic changes. These changes modify how genes are expressed and how cells function. The investigators want to study these epigenetic changes and the effect on peritoneal membrane scarring, blood vessel growth and peritoneal membrane function.

DETAILED DESCRIPTION:
There is considerable evidence that epigenetic changes in effector cells underlie the progressive nature of fibrogenic diseases. The investigators have developed an ex-vivo mesothelial cell culture system based on work by Aroeira and colleagues. Ex vivo cell cultures were treated with the DNA methyltransferase inhibitor 5-AZA for 72 hours. Overall, the investigators found that 11 of 14 patients' cells showed an increase in the E-Cad/alpha-SMA ratio with treatment to 5-AZA, indicating a return to a more epithelial-like phenotype and supporting an epigenetic mechanism of progressive fibrosis. The investigators hope to identify DNA methylation patterns associated with glucose exposure and peritoneal membrane solute transport in PD patients.

The investigators will take the peritoneal effluent from an overnight dwell from patients within one month of initiation of dialysis. The overnight effluent is centrifuged and the pellet is washed and cells are grown in DMEM medium. At confluence, cells are passaged into 2 flasks then taken for DNA and RNA. At 12 months, a second overnight peritoneal effluent sample will be obtained. The investigators will also gather demographic data (patient's age, diabetes, occurrence of peritonitis, cumulative PD prescription including total glucose exposure, use of icodextrin, and the results of a peritoneal equilibrium test carried out for clinical purposes between 3 and 12 months from the start of peritoneal dialysis). The investigators will use whole genome DNA methylation analysis to assess epigenetic changes in mesothelial cells from incident PD patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with end stage renal disease recently started on peritoneal dialysis. Patients will be over the age of 18.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with end stage renal disease recently started on peritoneal dialysis. Patients will be over the age of 18.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2015-09; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
DNA methylation pattern | 12 months
  DNA methylation pattern will be measured after 12 months of glucose exposure compared with a baseline sample. Gene expression will be measured by Genome wide methylation analysis. In the incident patients, a within-subject analysis will be carried out between the naive and 12 month cell culture sample. Gene expression analysis will be performed with the statistical software R and "BioConductor", a collection of tools for gene expression analysis. Gene-level summaries from Human HT-12 BeadChip data will be generated using the widely used Bioconductor package lumi, which includes background correction, variance stabilization and normalization of expression data. The Linear Models for Microarray Analysis (LIMMA) package of Bioconductor will be used for differential expression analysis.

SECONDARY OUTCOMES:
DNA methylation and solute transport | 12 months
  The investigators will correlate changes in DNA methylation with solute transport measured by a peritoneal equilibrium test and peritoneal glucose exposure. Solute transport is calculated from the dialysate to plasma creatinine ratio which is obtained from the peritoneal equilibrium test.

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Margetts, MD PhD, Principal Investigator — McMaster University
Locations (1):
- St. Joseph's Healthcare, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No